# Version 1.1 Version date 9/10/2020

# CONSENT BY PATIENT FOR CLINICAL RESEARCH

| I, |
|---|
| of |
| (Address) hereby agree to take part in the clinical research (clinical study/questionnaire study/drug trial) specified below: |
| <u>Title of Study:</u> The Immediate Effect of Mindfulness-Based Supportive Therapy (MBST) vs Supportive |
| Listening on Palliating Suffering in Palliative Care Cancer Patients: A Randomised Controlled Trial |
| the nature and purpose of which has been explained to me by Dr |
| and interpreted by |
| (Name & Designation of Interpreter) |
| to the best of his/her ability inlanguage/dialect. |
| I have been told about the nature of the clinical research in terms of methodology, possible adverse effects and complications (as per patient information sheet). After knowing and understanding all the possible advantages and disadvantages of this clinical research, I voluntarily consent of my own free will to participate in the clinical research specified above. |
| I understand that I can withdraw from this clinical research at any time without assigning any reason whatsoever and in such a situation shall not be denied the benefits of usual treatment by the attending doctors. |
| Date: |
| IN THE PRESENCE OF |
| Name) |
| Identity Card No. Signature |
| (Witness for Signature of Patient) |
| Designation) |
| I confirm that I have explained to the patient the nature and purpose of the above-mentioned clinical research. |
| Date |

CONSENT BY PATIENT FOR CLINICAL RESEARCH

R.N. Name Sex Age Unit

BK-MIS-1117-

# Version 1.1 Version date 9/10/2020

# KEIZINAN OLEH PESAKIT UNTUK PENYELIDIKAN KLINIKAL

| Saya, |
|---|
| beralamat(Alamat) |
| dengan ini bersetuju menyertai dalam penyelidikan klinikal (pengajian klinikal/pengajian soal-selidik/percubaan ubat-ubatan) disebut berikut: |
| <u>Tajuk Penyelidikan</u> : Keberkesanan terapi sokongan berasaskan latihan minda dalam mengurangkan sengsara di kalangan pesakit kanser. |
| yang mana sifat dan tujuannya telah diterangkan kepada saya oleh<br>Dr(Nama & Jawatan Doktor) |
| mengikut terjemahan |
| yang telah menterjemahkan kepada saya dengan sepenuh kemampuan dan kebolehannya di dalam Bahasa / loghat |
| Saya telah diberitahu bahawa dasar penyelidikan klinikal dalam keadaan methodologi, risiko dan komplikasi (mengikut kertas maklumat pesakit). Selepas mengetahui dan memahami semua kemungkinan kebaikan dan keburukan penyelidikan klinikal ini, saya merelakan/mengizinkan sendiri menyertai penyelidikan klinikal tersebut di atas. |
| Saya faham bahawa saya boleh menarik diri dari penyelidikan klinikal ini pada bila-bila masa tanpa memberi sebarang alasan dalam situasi ini dan tidak akan dikecualikan dari kemudahan rawatan dari doktor yang merawat. |
| Tarikh: |
| Nama) |
| No. K/P |
| ) (Saksi untuk Tandatangan Pesakit)<br>Jawatan) |
| Saya sahkan bahawa saya telah menerangkan kepada pesakit sifat dan tujuan penyelidikan klinikal tersebut di atas. |
| Tarikh: Tandatangan |

KEIZINAN OLEH PESAKIT
UNTUK
Jantina
PENYELIDIKAN KLINIKAL
Umur
Unit

BK-MIS-1117-E02

# CONSENT BY RESPONSIBLE RELATIVE FOR CLINICAL RESEARCH

| I, |
|---|
| of(Address) |
| hereby agree that my relative |
| I.C. No(Name) |
| participate in the clinical research (clinical study/questionnaire study/drug trial) specified below:- |
| Title of Study: The Immediate Effect of Mindfulness-Based Supportive Therapy (MBST) vs Supportive |
| Listening on Palliating Suffering in Palliative Care Cancer Patients: A Randomised Controlled Trial |
| the nature and purpose of which has been explained to me by Dr. |
| (Name & Designation of Doctor) |
| and interpreted by(Name & Designation of Interpreter) |
| to the best of his/her ability in language/dialect. |
| I have been informed of the nature of this clinical research in terms of procedure, possible adverse effects and complications (as per patient information sheet). I understand the possible advantages and disadvantages of participating in this research. I voluntarily give my consent for my relative to participate in this research specified above. |
| I understand that I can withdraw my relative from this clinical research at any time without assigning any reason whatsoever and in such situation, my relative shall not be denied the benefits of usual treatment by the attending doctors. Should my relative regains his/her ability to consent, he/she will have the right to remain in this research or may choose to withdraw. |
| Relationship Signature or Date: Thumbprint |
| IN THE PRESENCE OF |
| Name) |
| Identity Card No |
| Designation |
| I confirm that I have explained to the patient's relative the nature and purpose of the above-mentioned clinical research. |
| Date Signature |
| (Attending Doctor) |

### Version 1.1 Version date 9/10/2020

CONSENT BY Name
RESPONSIBLE RELATIVE FOR
CLINICAL RESEARCH Age
Unit

BK-MIS-1117-E02

### KEIZINAN OLEH WARIS YANG BERTANGGUNGJAWAB UNTUK PENYELIDIKAN KLINIKAL

| Saya, |
|---|
| beralamat(Alamat) |
| dengan ini bersetuju supaya saudara saya |
| dalam penyelidikan klinikal (pengajian klinikal/pengajian soal-selidik/percubaan ubat-ubatan) disebut berikut: |
| <u>TajukPenyelidikan:</u> Keberkesanan terapi sokongan berasaskan latihan minda dalam mengurangkan sengsara di kalangan pesakit kanser. |
| yang mana sifat dan tujuannya telah diterangkan kepada saya oleh Dr |
| (Nama & Jawatan Doktor) |
| mengikutterjemahan |
| (Nama & Jawatan Penterjemah) |
| yang telah menterjemahkan kepada saya dengan sepenuh kemampuan dan |
| kebolehannya di dalam Bahasa / loghat |
| Saya telah diberitahu bahawa dasar penyelidikan klinikal dalam keadaan metodologi, risiko dan komplikasi (mengikut kertas maklumat pesakit). Saya mengetahui dan memahami semua kemungkinan kebaikan dan keburukan penyelidikan klinikal ini. Saya merelakan/mengizinkan saudara saya menyertai penyelidikan klinikal tersebut di atas. |
| Saya faham bahawa saya boleh menarik balik penyertaan saudara saya dalam penyelidikan klinikal ini pada bilabila masa tanpa memberi sebarang alasan dalam situasi ini dan tidak akan dikecualikan dari kemudahan rawatan dari doktor yang merawat. Sekiranya saudara saya kembali berupaya untuk memberi keizinan, beliau mempunyai hak untuk terus menyertai kajian ini atau memilih untuk menarik diri. |
| Tarikh: Pertalian Tandatangan/Cap Jari Waris dengan Pesakit yang bertanggungjawab |
| DI HADAPAN |
| Nama) |
| No. K/P |
| Jawatan |
| Saya sahkan bahawa saya telah menerangkan kepada waris yang bertanggungjawab sifat dan tujuan penyelidikan klinikal tersebut di atas. |
| Tarikh: Tandatangan |
| (Doktor yang merawat) |
| No. Pend. |

KEIZINAN OLEH WARIS PESAKIT UNTUK PENYELIDIKAN KLINIKAL No. Pend Nama Jantina Umur Unit